CLINICAL TRIAL: NCT02798523
Title: Genomic Response of Human Immune and Non-Immune Cells to Glucocorticoids
Brief Title: Genomic Responses of Human Immune and Non-Immune Cells to Glucocorticoids
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 160126; 16-I-0126
Record Dates: First submitted 2016-06-10; First posted 2016-06-14 (Estimated); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2022-11-14

CONDITIONS: Normal Physiology
Keywords: Methylprednisolone; Immunologic; Glucocorticoids; Functional genomics; RNA; Steroids
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Up to 2 hours post infusion (Experimental): Healthy volunteers received a single intravenous dose of 250 mg of methylprednisolone and blood was collected between one to two hours after the start of the infusion.
  Interventions: Drug: Methylprednisolone sodium succinate(Solu-Medrol)
- Up to 4 hours post infusion (Experimental): Healthy volunteers received a single intravenous dose of 250 mg of methylprednisolone and blood was collected between two hours to four hours after the start of the infusion.
  Interventions: Drug: Methylprednisolone sodium succinate(Solu-Medrol); Drug: Topical methylprednisolone (Advantan emulsion 0 /1%)

INTERVENTIONS:
Drug: Methylprednisolone sodium succinate(Solu-Medrol) — Methylprednisolone sodium succinate for injection, USP (SOLU-MEDROL sterile powder, Pfizer, Inc.) is an anti-inflammatory glucocorticoid which occurs as a white, or nearly white, odorless hygroscopic, amorphous solid. It is very soluble in water and in alcohol; it is insoluble in chloroform and is very slightly soluble in acetone.
  125-milligram Act-O-Vial (AOV) System: Each 2 mL AOV (when mixed) contains methylprednisolone sodium succinate equivalent to 125 milligrams methylprednisolone; also 1.6 mg monobasic sodium phosphate anhydrous; and 17.4 mg dibasic sodium phosphate dried.
Drug: Topical methylprednisolone (Advantan emulsion 0 /1%) — 1 g Advantan emulsion 0.1% (Bayer) contains methylprednisolone aceponate (21-acetoxy-11beta-hydroxy-6alpha-methyl-17-propionyloxy-1,4-pregnadiene-3,20-dione) 1 mg, as the active ingredient. It is an oil-in-water emulsion containing medium chain triglycerides, caprylic-capric-stearic triglyceride, polyoxyethylene alcohol 2-stearyl ether, polyoxyethylene alcohol-21-stearyl ether, benzyl alcohol, disodium edetate, glycerol, and purified water.
  Arms: Up to 4 hours post infusion

SUMMARY:
Background:

The immune system defends the body against bacteria and other harmful invaders. But it can overact and attack healthy cells by mistake. The group of drugs called glucocorticoids (GCs) can calm down an overactive immune system. But they often cause negative side effects. Researchers want to learn how human genes respond to GCs. Genes live inside each cell of the body. They tell our cells how to function. Researchers hope the results of this study will show them how to develop better drugs that will have the benefits of GCs without the side effects.

Objectives:

To study how human genes respond to glucocorticoid drugs.

Eligibility:

Healthy adult volunteers ages 18-64.

Design:

Participants will be screened with a medical history and physical exam. They will have a heart test and blood tests.

The study visit will last about 6 hours.

Participants will have medical history, physical exam, and 3 blood draws.

Participants will have a skin biopsy. An injection will numb the skin on one arm. Then a tool will remove a piece of skin about as big as a pencil eraser.

A GC cream will be applied to the other arm.

Participants will get the GC study drug for 30 minutes. It will be a liquid that will drip through a needle placed in an arm vein.

Participants will have a skin biopsy of the arm that had the cream applied.

Participants will have follow-up calls 1 and 4 days later. They will be asked about reactions or other health problems.

DETAILED DESCRIPTION:
Glucocorticoids are among the most frequently prescribed immunosuppressive and anti-inflammatory medications worldwide. Long-term use, however, is complicated by serious non-immunologic side effects. Ongoing in vitro experiments with human primary cells in our laboratory suggest that there are indeed fundamental differences in the genomic response of immune and non-immune cells to glucocorticoids. These and other aspects of drug action at the genomic level have not been completely characterized. This study will attempt to generate a list of human genes and non-coding RNAs that are differentially expressed and regulated in response to glucocorticoids between immune and non-immune cells. These data will be used to identify transcripts, their corresponding proteins, and the molecular pathways that are best candidates for targeted intervention. Potential targets could be validated with small interfering RNA (siRNA) libraries, with the long-term goal of developing small-molecule or nanoparticle-facilitated RNA interference (RNAi) interventions that reproduce the therapeutic action of glucocorticoids in immune cells while avoiding their harmful side effects on other tissues.

Healthy volunteers will undergo baseline blood collection prior to receiving a single intravenous dose of 250 milligrams of methylprednisolone sodium succinate. Blood will be collected in one of two regimens: 1 and 2 hours or 2 and 4 hours after the start of the infusion. A skin punch biopsy may be obtained before healthy volunteers receive IV methylprednisolone. If so, topical methylprednisolone will be applied to a limited area of skin, contralateral to the site of the baseline skin biopsy, and an additional skin biopsy will be obtained 4 hours after drug administration, from the area where topical methylprednisolone was applied. Follow-up phone calls 1 day and 1 week after discharge will document any adverse effects related to the drug or skin biopsy. Total length of individual study participation is 1-5 weeks.

Blood samples will be processed for isolation of hematopoietic cell sub-population (neutrophils, B cells, CD4+ T cells, CD8+ T cells, monocytes, and natural killer [NK] cells). Laboratory studies will be performed in the purified cells, with the goal of understanding the human response to glucocorticoids in vivo at the level of RNA (e.g., RNA sequencing, small -RNA-sequencing, real-time PCR), DNA (e.g., ChIP-seq, methylation analysis, DNA sequencing, genotyping, and protein (e.g., flow cytometry, mass spectrometry). At each time point, serum methylprednisolone levels will be measured and flow cytometry for standard lineage markers will be performed. Skin biopsies will be subjected to RNA isolation for RNA sequencing and small-RNA sequencing. A fragment of each skin biopsy will undergo fibroblast isolation and culture for in vitro exposure to glucocorticoids and for the generation of induced pluripotent stem (iPS) cells.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 18 to 64 years
  2. Willingness to have samples stored for future research
  3. Willingness to undergo genetic testing

EXCLUSION CRITERIA:

1. Body Mass Index less than 18 or greater than 35
2. Difficult peripheral venous access (as determined by study staff at screening)
3. History of severe allergic reaction to glucocorticoids
4. History of autoimmune or autoinflammatory disease
5. Active solid or hematologic malignancy
6. History of a skin condition (such as psoriasis, pemphigus, or atopic dermatitis) that could affect the results of the transcriptional analysis of the skin biopsy samples
7. Diabetes mellitus
8. Cancer chemotherapy within the past 5 years
9. Surgery within the past 8 weeks
10. History of recent (within the past 30 days) infection
11. A positive test for human immunodeficiency virus, or hepatitis A, B or C virus infection (viral markers hepatitis screen, which includes HBsAg, anti-HCV IgG, anti-HAV IgM).
12. A positive or indeterminate test for latent tuberculosis (interferon gamma release assay)
13. History of parasitic, amebic, fungal or mycobacterial infections, or other possible latent infections
14. Coagulation test (PT and PTT) results outside of normal range
15. History of a bleeding disorder
16. Use of a glucocorticoid (including topical or inhaled), a nonsteroidal anti-inflammatory drug (including aspirin), an anti-epileptic drug, an anticoagulant, a statin, fluoxetine, diltiazem, amiodarone, clarithromycin, ketoconazole, or St. John s wort, within the past 30 days
17. Vaccination within the past 30 days
18. Receipt of an immunosuppressant or immunomodulatory drug within the past 30 days
19. Pregnancy, current or within the past 90 days, or trying to become pregnant during the study
20. Current breastfeeding
21. Complete blood count (CBC) and/or acute care panel values are both outside of the NIH Department of Laboratory Medicine normal reference range and deemed clinically significant by the principal investigator
22. Any Electrocardiogram (ECG) abnormality that is clinically significant
23. Any condition that, in the investigator s opinion, may put the participant at undue risk or compromise the study s scientific objectives
24. Participation in a clinical protocol which includes an intervention that, in the opinion of the investigator, may affect the results of the current study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis M Franco, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Khoury P, Stokes K, Gadkari M, Makiya MA, Legrand F, Hu Z, Klion A, Franco LM. Glucocorticoid-induced eosinopenia in humans can be linked to early transcriptional events. Allergy. 2018 Oct;73(10):2076-2079. doi: 10.1111/all.13497. Epub 2018 Jul 17. No abstract available. PMID 29885264
- [Background] Franco LM, Gadkari M, Howe KN, Sun J, Kardava L, Kumar P, Kumari S, Hu Z, Fraser IDC, Moir S, Tsang JS, Germain RN. Immune regulation by glucocorticoids can be linked to cell type-dependent transcriptional responses. J Exp Med. 2019 Feb 4;216(2):384-406. doi: 10.1084/jem.20180595. Epub 2019 Jan 23. PMID 30674564
- [Background] Gadkari M, Makiya MA, Legrand F, Stokes K, Brown T, Howe K, Khoury P, Hu Z, Klion A, Franco LM. Transcript- and protein-level analyses of the response of human eosinophils to glucocorticoids. Sci Data. 2018 Dec 4;5:180275. doi: 10.1038/sdata.2018.275. PMID 30512017
- [Derived] Hong SG, Sato N, Legrand F, Gadkari M, Makiya M, Stokes K, Howe KN, Yu SJ, Linde NS, Clevenger RR, Hunt T, Hu Z, Choyke PL, Dunbar CE, Klion AD, Franco LM. Glucocorticoid-induced eosinopenia results from CXCR4-dependent bone marrow migration. Blood. 2020 Dec 3;136(23):2667-2678. doi: 10.1182/blood.2020005161. PMID 32659786
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-I-0126.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 33 subjects who consented to the protocol, eight subjects were screen failure and 25 unique subjects participated in the study. One subject participated in both arms of the study
Period: 2 Hour or 4 Hour Post Infusion
Arm/Group | Up to 2 Hours Post Infusion | Up to 4 Hours Post Infusion
Started | 4 | 21
Completed | 4 | 21
Not Completed | 0 | 0
Period: 4 Hours Then 2 Hours Post Infusion
Arm/Group | Up to 2 Hours Post Infusion | Up to 4 Hours Post Infusion
Started | 0 | 1 (One subject from the 4-hour post infusion arm also participated in the 2-hour post infusion arm)
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Up to 2 Hours Post Infusion | Up to 4 Hours Post Infusion | Total
Number analyzed (Participants) | 4 | 21 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 21 | 25
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 10 | 12
  Male | 2 | 11 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 3 | 17 | 20
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 3 | 13 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Sampled for RNA-seq Differential Expression Analysis (Biological Replicates)
Description: Number of participants (biological replicates) that were successfully sampled for RNA-seq differential gene expression analysis in glucocorticoid-treated immune cells. The analysis employed a cutoff value of < 5% false-discovery rate (FDR) to select the transcripts that were considered differentially expressed at each time point. The resulting gene lists were contrasted to determine which genes were uniquely differentially expressed in different cell types.
Time Frame: Up to 2 or 4 hours post infusion depending on group
Population: Participants who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Up to 2 Hours Post Infusion | Up to 4 Hours Post Infusion
Number analyzed (Participants) | 5 | 21
Participants | 5 | 20

ADVERSE EVENTS:
Time Frame: Up to five days
Arm/Group | Up to 2 Hours Post Infusion | Up to 4 Hours Post Infusion
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/21
Other Adverse Events (participants affected / at risk) | 2/5 | 16/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Up to 2 Hours Post Infusion (N=5) | Up to 4 Hours Post Infusion (N=21)
Palpitations (Cardiac disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Application site pain (General disorders) | 0 | 1
Application site pruritus (General disorders) | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 2
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 6
Presyncope (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Sleep disorder (Psychiatric disorders) | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT02798523/Prot_SAP_000.pdf